CLINICAL TRIAL: NCT03333850
Title: Technology Assisted Physical Activity Among Hospitalised Patients With Respiratory Disease - a Controlled Cohort Study
Brief Title: Technology Assisted Physical Activity Among Hospitalised Patients With Respiratory Disease
Acronym: TAPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: FYS010
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: There will be sequential inclusion to each cohort. Each sequence includes 18 patients (corresponding to the number of beds at the department). Thus the patients hospitalised during the first period will receive feedback (exposed cohort). In the second period the patients will not receive feedback (non-exposed cohort), and so forth. A total of 108 patients will be included resulting in 6 periods of 18 patients each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual feedback of physical activity (Experimental): Participants in the exposure cohort will receive usual hospital care and continuous measurement of physical activity by sensors collecting physical activity level during hospitalisation AND a monitor placed at their bedside that displays information about their physical activity level, in terms of time spent bedridden, sitting, standing and walking. This information will be visible to the health personnel, the patients and their relatives.
  Interventions: Device: Visual feedback of physical activity; Device: Measurement of physical activity
- No feedback of physical activity (Active Comparator): The participants in the non-exposure cohort will receive usual hospital care and continuous measurement of physical activity by sensors collecting physical activity level during hospitalisation. No visual feedback is provided.
  Interventions: Device: No feedback of physical activity; Device: Measurement of physical activity

INTERVENTIONS:
Device: Visual feedback of physical activity — A monitor (tablet) will display the level of physical activity during hospitalisation. The monitor will be placed at the bedside (table).
  Arms: Visual feedback of physical activity
Device: No feedback of physical activity — There will be no visual feedback of the physical activity (no monitor placed at the bedside (table)).
  Arms: No feedback of physical activity
Device: Measurement of physical activity — A pair of accelerometers placed on the chest and on the thigh will measure the physical activity level during hospitalisation. The measurement is made continuously and stored on a secure web-server.

SUMMARY:
The aim of this study is to investigate if patients hospitalised for medical disease will increase their time spent out of bed during hospitalisation through simple feedback about physical activities from a mobile device.

Physical activity is measured by means of a pair of accelerometers embedded in band aids placed on the thigh and on the chest. The measurement is continuous and data is uploaded to a secure internet-server. Summaries of physical activity (bedrest, sitting, standing, walking) is computed and can be displayed on a mobile device (tablet) through a dedicated application.

The study will be conducted as a controlled cohort study in a large tertiary public hospital in Copenhagen, Denmark. Patients admitted to Department of Respiratory Medicine will be included and will have their physical activity measured during hospitalisation. Half of the cohort will receive visual feedback about the amount of physical activity from a mobile device placed on the bed table.

A total of 108 patients will be included resulting in 6 periods of 18 patients each.

ELIGIBILITY:
Inclusion Criteria:

1. Is admitted to the Department of Respiratory Medicine
2. Has signed informed consent
3. Reads and speaks Danish

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator, makes the person unfit for participation
2. Has allergy towards band aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Time spent out of bed during hospitalisation | 7 Days
  Time (in minutes) spent out of bed measured in minutes related to the total hospitalisation time. The time spent out of bed will be recorded throughout the hospitalisation for a maximum of 7 days.

SECONDARY OUTCOMES:
Time spent sitting during hospitalisation | 7 Days
  Time (in minutes) spent sitting related to the total hospitalisation time. The time sitting will be recorded throughout the hospitalisation for a maximum of 7 days.
Time spent standing during hospitalisation | 7 Days
  Time (in minutes) spent standing related to the total hospitalisation time. The time standing will be recorded throughout the hospitalisation for a maximum of 7 days.
Time spent walking during hospitalisation | 7 Days
  Time (in minutes) spent walking related to the total hospitalisation time. The time walking will be recorded throughout the hospitalisation for a maximum of 7 days.

OTHER OUTCOMES:
Mortality | 7 Days
  Mortality at any time during hospitalisation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Dall, PhD, Study Director — Department of Physio- and Occupational Therapy, Bispebjerg-Frederiksberg Hospital, Denmark; Marius Henriksen, PhD, Principal Investigator — Department of Physio- and Occupational Therapy, Bispebjerg-Frederiksberg Hospital, Denmark
Locations (1):
- Bispebjerg Hospital, Department of Physical and Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
When data has been anonymised, analysed, and the scientific report(s) published, the data will be made available to other researchers. Availability will be through direct contact to the study director or principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When data has been anonymised, analysed, and the scientific report(s) published.
Access Criteria: The are no criteria specified at this time